CLINICAL TRIAL: NCT02710357
Title: Single-implant Mandibular Overdenture or a Conventional Complete Denture? A Cost-effectiveness Analysis Alongside a Randomized Clinical Trial
Brief Title: A Cost-effectiveness Analysis of the Single-implant Mandibular Overdenture Treatment
Acronym: SIMOECON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Principal Investigator, Cláudio Rodrigues Leles, Associate professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 966_2014
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Mouth, Edentulous
Keywords: Mandibular Prosthesis Implantation; Prostheses and Implants; Denture, Complete, Lower
MeSH Terms: conditions — Mouth, Edentulous | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mandibular complete denture (Active Comparator): Participants allocated to this group will not receive any additional treatment. When needed, retreatment or any adjustment/repair in the dentures will be performed accordingly. Participants will receive regular maintenance for their dentures, including adjustments for the elimination of sore areas, denture relining and repair of fractures, when needed, until the end of the follow-up period.
  Interventions: Procedure: Mandibular complete denture
- Single-implant mandibular overdenture (Experimental): Participants allocated to this group will have an implant placed in the mandibular midline and after 4 weeks (healing period - early loading) an attachment system will be tightened and a retention matrix will be incorporated to the mandibular denture.
  Interventions: Procedure: Mandibular Overdenture

INTERVENTIONS:
Procedure: Mandibular Overdenture — Placement of an implant in the mandibular midline.
  Other Names: Dental Implant (Straumann Standard Plus SLActive® RN implant
  Arms: Single-implant mandibular overdenture
Procedure: Mandibular complete denture — No intervention. Maintenance of the dentures will be done when needed.
  Arms: Mandibular complete denture

SUMMARY:
The aim of this study is to assess the cost-effectiveness of the mandibular overdenture retained by a single implant. The study hypothesis is that SIMO is more effective but more costly than the conventional denture, though this incremental cost is relatively low for the offered effectiveness in terms of clinical and patient-reported outcomes.

DETAILED DESCRIPTION:
This randomized clinical trial alongside a cost-effectiveness analysis will include twenty-eight edentulous individuals who meet eligibility criteria. New maxillary and mandibular dentures will be fabricated for all participants following a standardized protocol. Then, participants will be randomized into one of the treatment groups: conventional complete denture group or single-implant mandibular overdenture group. Each participant allocated to the overdenture group will then receive a Straumann® Standard Plus SLActive® regular neck implant (Straumann 0.33.051S/052S/053S Institute Straumann AG, Basel, Switzerland) in the mandibular midline. A healing abutment will be connected and the implant will be allowed to heal for approximately 3 weeks. Then, a 3.4mm retentive titanium anchor abutment (Straumann 048.439, Institute Straumann AG, Basel, Switzerland) will be connected and tightened to 35 N.cm with a torque wrench. The matrix will be incorporated to the denture using self-curing acrylic resin and the patient will be instructed to keep the upper and lower dentures firmly occluded in the habitual position until the final polymerization of the resin. Direct costs related to therapies in both groups will be identified, measured and valuated for one year after treatment and patient-reported outcomes will be assessed. Incremental cost-effectiveness ratios will be estimated and graphically presented on cost-effectiveness planes. A Markov decision tree will be constructed to set out the consequences of the competing alternatives. Sensitivity analysis on the most important assumptions will be performed in order to assess the robustness of the model.

ELIGIBILITY:
Inclusion Criteria:

* No contraindications for implant surgery (mainly related to uncontrolled systemic diseases)
* Present enough bone volume in the mandibular midline area for implant placement without the need of bone augmentation procedures.
* Be able to understand and answer the questionnaires used in the study
* Agree to participate by providing a written informed consent.

Exclusion Criteria:

* Noncompliant participants
* Individuals who do not agree to be randomly allocated to the treatment study group
* Presence of signs of untreated temporomandibular disorders, uncontrolled systemic or oral conditions that require additional treatments

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Oral health-related quality of life impacts | Changes from baseline to 12 months after the intervention
  The cross-culturally adapted Brazilian version of the Oral Health Impact Profile for edentulous subjects (OHIP-EDENT) will be used. It contains 19 items divided in four different subscale domains: (I) masticatory discomfort and disability (four items), (II) psychological discomfort and disability (five items), (III) social disability (five items), and (IV) oral pain and discomfort (five items). The items are answerable by a 3-point Likert scale and responses will be summed to result an overall score. Higher scores represent worse OHRQoL.
Satisfaction with the dentures | Changes from baseline to 12 months after the intervention
  A 10 cm uninterrupted visual analogue scale will be used in order to assess the participants' ratings of their satisfaction with the upper and lower dentures in relation to the parameters "general satisfaction", "comfort", "stability", "aesthetics", "ability to speak" and "ability to chew". Each participant will indicate their level of satisfaction with each parameter by marking a point along the scale, in which ends mean "unsatisfied" and "satisfied", as it is closer to the beginning or the end of the scale, respectively.

SECONDARY OUTCOMES:
Masticatory efficiency | Changes from baseline to 12 months after the intervention
  Masticatory efficiency will be assessed as a secondary outcome using a two-colored chewing gum test and a qualitative and quantitative colourimetric method to measure the color-mixing ability. Participants will be asked to sit upright in a dental chair and to chew the gum on their preferred chewing side for 20 cycles. Visual and electronic analysis of the chewed gums samples will be done according to the classification proposed by Schimmel et al. Analysis will be made by two investigators blinded to the study groups and treatment stage. The software ViewGum (dHAL Software, Kifissia, Greece, www.dhal.com) will be used for electronic colourimetric analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio R Leles, DDS, PhD, Study Director — Universidade Federal de Goias
Locations (1):
- School of Dentistry, Federal University of Goias, Goiânia, Goiás, Brazil

REFERENCES:
- [Derived] Nogueira TE, Esfandiari S, Leles CR. Cost-effectiveness analysis of the single-implant mandibular overdenture versus conventional complete denture: study protocol for a randomized controlled trial. Trials. 2016 Nov 4;17(1):533. doi: 10.1186/s13063-016-1646-0. PMID 27814749